CLINICAL TRIAL: NCT07026799
Title: Investigation of an Exercise Intervention for Multiple Myeloma Patients With Stable and Unstable Osteolytic Lesions During Induction Therapy.
Brief Title: Feasibility, Safety and Effectivity of an Exercise Intervention for Newly Diagnosed Multiple Myeloma Patients During Induction Therapy
Acronym: GMMG-HD8-INDEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Ulrike Dapunt, Prof. Dr. med., University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-165/2023
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma Bone Lesions
Keywords: orthopaedic evaluation of bone stability; Multiple myeloma; Physical exercise; Osteolysis
MeSH Terms: conditions — Multiple Myeloma; Motor Activity; Osteolysis | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator)
  Interventions: Other: Exercise
- Control group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Exercise — Orthopedic consultation and home-based, individualized, structured resistance training during induction therapy.
  Arms: Intervention group
Other: Control group — Orthopedic consultation and stretching exercises/walking. No resistance training.
  Arms: Control group

SUMMARY:
Physical exercise is an important supportive therapy for cancer patients, which improves quality of life and can effectively counteract the side effects of drug therapy. There is very little experience whether physical activity can also be performed safely by patients with malignant diseases that affect bone stability. This applies in particular to patients with multiple myeloma, a disease characterized by a monoclonal proliferation of plasma cells in the bone marrow and often accompanied by severe bony destruction. Aim of this exploratory randomized controlled trial is to evaluate feasibility, safety and effectivity of an orthopaedic-guided exercise intervention during induction therapy in newly diagnosed multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed multiple myeloma
* Survival prognosis > 6 months
* ECOG status ≤ 3
* Age ≥18 years
* Patients who state that they want to carry out the training program at least 2 x/week and participate in the planned follow-up visits
* Ability to give informed consent
* Written consent to participate in the study
* Sufficient knowledge of written and spoken German

Exclusion Criteria:

* physical or mental limitation that would prevent participation in the training program or the planned follow-up visits.
* Carrying out a regular, intensive training program (min. 1h, 2x/week)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Fatigue (MFI, Multidimensional Fatigue Inventory) | From enrollment to the end of stem cell transplantation (approximately one year)

CONTACTS AND LOCATIONS:
Locations (1):
- Heidelberg University Hospital - GMMG Study Group, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
* questionnaire results collected for each individual
  * functional test results collected for each individual

REFERENCES:
- [Background] Courneya KS, Vardy JL, O'Callaghan CJ, Gill S, Friedenreich CM, Wong RKS, Dhillon HM, Coyle V, Chua NS, Jonker DJ, Beale PJ, Haider K, Tang PA, Bonaventura T, Wong R, Lim HJ, Burge ME, Hubay S, Sanatani M, Campbell KL, Arthuso FZ, Turner J, Meyer RM, Brundage M, O'Brien P, Tu D, Booth CM; CHALLENGE Investigators. Structured Exercise after Adjuvant Chemotherapy for Colon Cancer. N Engl J Med. 2025 Jul 3;393(1):13-25. doi: 10.1056/NEJMoa2502760. Epub 2025 Jun 1. PMID 40450658
- [Background] Nicol JL, Woodrow C, Burton NW, Mollee P, Nicol AJ, Hill MM, Skinner TL. Physical Activity in People with Multiple Myeloma: Associated Factors and Exercise Program Preferences. J Clin Med. 2020 Oct 13;9(10):3277. doi: 10.3390/jcm9103277. PMID 33066153
- [Background] Nicol JL, Hill MM, Burton NW, Skinner TL. Promoting exercise for patients with multiple myeloma: attitudes and practices of clinical haematologists. J Cancer Surviv. 2022 Jun;16(3):688-695. doi: 10.1007/s11764-021-01062-2. Epub 2021 Jun 11. PMID 34114194
- [Background] Bower JE. Cancer-related fatigue--mechanisms, risk factors, and treatments. Nat Rev Clin Oncol. 2014 Oct;11(10):597-609. doi: 10.1038/nrclinonc.2014.127. Epub 2014 Aug 12. PMID 25113839
- [Background] Christensen JF, Simonsen C, Hojman P. Exercise Training in Cancer Control and Treatment. Compr Physiol. 2018 Dec 13;9(1):165-205. doi: 10.1002/cphy.c180016. PMID 30549018